CLINICAL TRIAL: NCT00553943
Title: Prospective Multicentre Phase II Study to Evaluate the Combination of Rituximab and DepoCyte® by Intrathecal Injection in the C5R Chemotherapy Protocol in Patients Between the Ages of 18 and 60 Years With Primary Cerebral Non-Hodgkin Lymphoma and Systemic Diffuse Large B-cell Lymphoma With Neuromeningeal Invasion at Diagnosis
Brief Title: Phase II Study to Evaluate the Combination of Rituximab and DepoCyte® in the C5R Chemotherapy Protocol in Patients Between the Ages of 18 and 60 Years With Primary Cerebral Non-Hodgkin Lymphoma and Systemic Diffuse Large B-cell Lymphoma With Neuromeningeal Invasion at Diagnosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-C5R 2006
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Lymphoma, Non-Hodgkin; Diffuse Large B-cell Lymphoma
Keywords: lymphoma; cerebral lymphoma; central nervous system; cytarabine; rituximab; Diffuse large B-cell lymphomas, with cerebral or neuromeningeal involvement
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma; Dendritic Cell Sarcoma, Interdigitating | interventions — Rituximab; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rituximab + Cytarabine (Experimental)
  Interventions: Drug: Rituximab; Drug: Cytarabine

INTERVENTIONS:
Drug: Rituximab — 375 mg/m2 D1
Drug: Cytarabine — 50 mg D3

SUMMARY:
The purpose of this study is to measure the rate of complete response (CR and UCR) at the end of a course of immuno-chemotherapy:

* before cerebral radiotherapy for PCL
* after the course of immuno-chemotherapy for aggressive lymphomas with neuromeningeal involvement Toxicity of the protocol Overall survival Survival without relapse Long-term incidence of neurocognitive toxicity

ELIGIBILITY:
Inclusion Criteria:

* Primary cerebral or oculocerebral NHL not previously treated with chemotherapy or radiotherapy and diffuse large B-cell lymphomas, with cerebral and / or neuromeningeal involvement at diagnosis.
* Diagnosis proved by histological or cytological examination of cerebral specimens, CSF or vitreous humour.
* Diffuse large cell CD20+ lymphoma.
* Men or women between the ages of 18 and 60 years.
* Presence of a measurable target to evaluate response.
* Negative serological tests for HIV, hepatitis B (except in cases of vaccination), hepatitis C.
* Life-expectancy ≥ 3 months
* Patient having given written consent to participate in this study.

Exclusion Criteria:

* CD20- lymphoma.
* History of indolent lymphoma, treated or untreated.
* Contraindication for one of the products used in polychemotherapy.
* Known hypersensitivity to mouse antibodies.
* Absence of measurable target to evaluate response.
* History of cancer in the 5 years prior to inclusion except for cutaneous basocellular carcinomas and non-invasive carcinomas of the neck of the uterus.
* Cardiac contraindication to treatment with anthracyclines or to hyperhydration:

SEVERE DISTURBANCE OF HEART RHYTHM VENTRICULAR EJECTION FRACTION BELOW 50% HISTORY OF RECENT MYOCARDIAL INFARCTION

* Previously known severe renal insufficiency and/or creatinaemia >150 µM/L (apart from invasion of the kidneys by the lymphoma).
* Total bilirubin >30 µmol/L, ASAT, ALAT >2.5 times the upper normal value (apart from invasion of the liver by the lymphoma).
* Insufficient medullary reserve: PNL < 1 G/L and platelets <100 G/L (apart from invasion of the medulla by the lymphoma).
* History of organ transplantation or other causes of severe immunosuppression.
* Pregnant woman.
* Patient incapable of keeping to regular monitoring.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2007-07 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Response to treatment (CR/PR) | End of treatment - 5 months

SECONDARY OUTCOMES:
Toxicity, Overall survival, Time to progression | End of study - 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Herve Ghesquieres, MD, Study Chair — LYmphoma Study Association (LYSA)
Locations (46):
- Belgium (11):
  - ZNA Stuivenberg, Antwerp
  - Hôpital Saint Joseph, Arlon
  - A. Z. Sint-Jan, Bruges
  - UCL- Saint Luc, Brussels
  - CH Notre Dame, Charleroi
  - AZ VUB, Jette
  - CHR de la Citadelle, Liège
  - CHU Charleroi-Vésale, Montigny-le-Tilleul
  - Clinique Saint Pierre, Ottignies
  - Heilig Hart Ziekenhuis, Roeselare
  - UCL - Mont-Godinne, Yvoir
- France (35):
  - CH d'Annecy, Annecy
  - Centre Hospitalier d'Avignon, Avignon
  - Hôpital de Bayonne, Bayonne
  - Hôpital d'Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - CH de Brive, Brive-la-Gaillarde
  - CHU Clemenceau, Caen
  - Centre Francois Baclesse, Caen
  - CH de Chambery, Chambéry
  - CH de Chartres, Chartres
  - Hôpital Gilles de Corbeil, Corbeil-Essonnes
  - Hôpital Henri Mondor, Créteil
  - CHU Le Bocage, Dijon
  - Centre Hospitalier de Dunkerque, Dunkirk
  - Hôpital Saint Louis, La Rochelle
  - Hôpital Andre Mignot, Le Chesnay
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Lens, Lens
  - Hopital Saint Vincent de Paul, Lille
  - CHU Claude Huriez, Lille
  - Hôpital Dupuytren, Limoges
  - Centre Leon Berard, Lyon
  - Hôpital des Chanaux, Mâcon
  - CH de Meaux, Meaux
  - Hôpital Bon Secours, Metz
  - Hôpital Emile Muller, Mulhouse
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint Louis, Paris
  - Hôpital Necker, Paris
  - Centre Hospitalier de Perpigan, Perpignan
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
  - CH de St Germain, Saint-Germain-en-Laye
  - Hôpital Purpan, Toulouse
  - Hopital Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.gela.org